CLINICAL TRIAL: NCT06686147
Title: Comparison of Range of Motion in Patients With Low Back Pain Using Artificial Intelligence-Assisted Analysis Method
Brief Title: AI-Assisted Analysis of Range of Motion in Patients With Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Seref Duhan Altug, M.Sc., Pamukkale University
Other Study IDs: Sltug
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Back Pain Patient Group
  Interventions: Diagnostic Test: Assessment of Joint Range of Motion
- Healthy Control Group
  Interventions: Diagnostic Test: Assessment of Joint Range of Motion

INTERVENTIONS:
Diagnostic Test: Assessment of Joint Range of Motion — Joint range of motion (ROM) measurements will be conducted to assess the specific ranges of motion of participants' joints.

SUMMARY:
Low back pain (LBP) is a common musculoskeletal problem that is frequently encountered in the population and can occur at any age. Responsible for the loss of a full healthy year in both the 10-24 and 50-74 age groups, LBP causes significant personal and social losses and increases healthcare costs.

In the classification of low back pain, pain that persists for up to 6 weeks is defined as acute, pain that lasts between 6-12 weeks is subacute, and pain that persists for more than 12 weeks is considered chronic low back pain (CLBP).

Chronic LBP (CLBP) leads to fear of movement, causing patients to limit their daily activities and social participation to avoid pain. A sedentary lifestyle in LBP patients is a factor that contributes to the chronicity of the disease. While most acute LBP patients recover well within a few weeks or months, the prognosis for patients with chronic low back pain is generally poor. Approximately one-quarter of patients visiting primary care facilities develop chronic LBP.

Therefore, identifying the risk factors for chronic LBP, understanding the population at risk of developing chronic LBP, identifying high-risk individuals, and implementing appropriate preventive and therapeutic measures are important.

Several musculoskeletal problems have played a role as risk factors in the development of LBP, and identifying and validating these risk factors can provide a potential mechanism through which LBP can be effectively treated. Accurately identifying musculoskeletal problems and risk factors can provide a mechanism to prevent the development of LBP and reduce the socioeconomic burden associated with the condition.

Machine learning (ML) is a scientific discipline that uses computer algorithms to identify patterns in large amounts of data and make predictions on new datasets based on these patterns. ML creates models to predict unknown data from historical data and allows us to select the most appropriate algorithm. Additionally, ML algorithms can extract variables that contribute to the prediction of the target variable, and differ from traditional statistical methods in enhancing the accuracy of future data predictions. ML has shown excellent performance in increasing the predictive value of medical imaging and postoperative clinical outcomes.

The aim of this study is to compare the joint range of motion in patients with low back pain and healthy individuals, and to detect differences in these ranges using artificial intelligence-supported analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Individuals who have experienced lower back pain for at least 3 months
* Individuals who have consulted a doctor at least once due to lower back pain
* Individuals who agree to participate in the study and have signed the informed consent form

Exclusion Criteria:

* Individuals who have undergone surgical intervention due to lower back pain
* Individuals with acute traumatic injuries
* Individuals with neurological or systemic diseases unrelated to the musculoskeletal system
* Individuals who have received physiotherapy or surgical treatment for lower back pain in the last three months
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic low back pain patient
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Evaluation | 5 minute
  This outcome measure assesses changes in pain levels using the Visual Analog Scale (VAS), a validated tool for pain evaluation. Pain intensity will be recorded by having participants rate their pain on a scale from 0 (no pain) to 10 (worst possible pain). Pain assessments will be conducted at baseline and follow-up intervals to track changes in reported pain intensity over time. The VAS provides a quantitative measurement of pain that is sensitive to minor changes, allowing for accurate monitoring of treatment effectiveness or condition progression.
Joint Range of Motion (ROM) | 20 minutes
  The primary outcome for this clinical study is the evaluation of Joint Range of Motion (ROM) in degrees (°), measured using the Halo digital goniometer. The assessment will include both active and passive ROM for major joints: shoulder, elbow, wrist, neck, lumbar spine, hip, knee, and ankle. Each joint's ROM will be recorded in degrees to provide a quantitative measure of flexibility and mobility. Data will be analyzed against normative values to determine any deviation or restriction in movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No